CLINICAL TRIAL: NCT05467020
Title: Association Between Peripheral Muscle Function and Quality of Life in Obese Subjects.
Acronym: OVALIA
Status: Completed | Type: Observational
Sponsor: Hopital Forcilles (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-A03248-33
Record Dates: First submitted 2022-07-15; First posted 2022-07-20 (Actual); Last update posted 2023-10-11 (Actual); Status verified 2022-07

CONDITIONS: Obesity
Keywords: obesity; muscle assessment; ultrasonography
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The assessment of health status and physical function is fundamental in patients with obesity, as they play an important role among the various factors influencing the quality of life in this population. Several studies have shown an association between high BMI values and a significant deterioration in quality of life, especially in women. Excess body fat in obese patients seems to be responsible for muscle atrophy. This causal link is probably related to dysfunctions in adipose tissue, leading to a decrease in the expression of proteins responsible for muscle contraction. The recent literature highlights an alteration in quality of life, particularly in obese and elderly subjects, for which changes in muscle function are partly responsible. Changes in muscle function can be assessed by simple, rapid and non-invasive tools. They could be used to identify obese subjects at risk of they could be used to identify obese subjects at risk of muscle atrophy, to stratify the risk, and to propose prophylactic intervention or early management.

The main objective of this study is to evaluate the association between structural alteration of the quadriceps and quality of life in obese patients.

The secondary objectives are to evaluate :

* The association between quadriceps thickness and quality of life ;
* The association between grip strength and quality of life ;
* The association between quadriceps strength and quality of life ;
* The association between quadriceps strength and ultrasound measurements of the quadriceps.

This is a prospective, monocenter, observationnal and cohort study.

All outpatients for nutrition assessment will be included.

DETAILED DESCRIPTION:
1. Rationale 1.1 Obesity, a global public health Obesity is a disease of multifactorial origin, linked to nutritional alterations, genetic, psychological, socio-economic factors and more sedentary behaviour (4) (5). The prevalence of obesity continues to increase in all age groups and in all socio-economic groups.

   1.2 Functional consequences of obesity. Patients with obesity with or without metabolic disorders have impaired health, including mental problems and reduced quality of life (12). In younger obese subjects the investigators also observe a decrease in quality of life compared to normal weight subjects, where muscle capacity may be a potential factor associated with impaired quality of life (13).

   1.2.1 Peripheral muscle damage A decrease in the specific force of the muscle, a decrease in force in relation to the sectional area, is observed in subjects with obesity. There is therefore probably a structural alteration of the muscle in the obese patient, which has not yet been described in the literature (17).

   1.3 Peripheral muscle ultrasound Muscle ultrasound measurements have become increasingly used as a non-invasive method of determining muscle characteristics (21). Muscle characteristics, particularly muscle size and quality, have been shown to be related to muscle strength and power as well as cardiovascular performance.
2. Research hypothesis The investigators hypothesise that impaired peripheral muscle function is associated with impaired quality of life in obese subjects.

3 Objective 3.1 Main objective The main objective of this study is to evaluate the association between structural alteration of the quadriceps and quality of life in obese patients.

3.2 Secondary objectives

The secondary objectives are to evaluate :

* The association between quadriceps thickness and quality of life ;
* The association between grip strength and quality of life ;
* The association between quadriceps strength and quality of life ;
* The association between quadriceps strength and ultrasound measurements of the quadriceps.

  4. Type of study This is a prospective, monocenter, obversational cohort study. The research will be conducted in accordance with the protocol.

  5. The duration of recruitment will be 9 months.

  6. Standard assessment procedures: Hand Grip Force, Maximum Voluntary Force of the quadriceps.

  7. Assessment procedures added by the research: Muscle ultrasound and Quality of Life Scale.

  8. Statistical aspects: Statistics will be primarily descriptive and will be based on means (+/- standard deviation) or medians [minimum-maximum] depending on the distribution of quantitative variables. Qualitative variables will be described in terms of numbers and percentages. Univariate comparisons will use the usual statistical tests after verification of the distribution of the variables (Chi2 or Fisher's test, t-test, anova or their non-parametric equivalents Wilcoxon and Kruskal-Wallis tests).

The risk of low quality of life in the presence of impaired muscle function will be described by the Odd-Ratios.

Tests will be performed at the 5% significance level. The 95% confidence intervals will be provided for each estimate.

9. Expected results in terms of scientific and professional advances: This study will evaluate the association between peripheral muscle function and quality of life impairment in obese patients hospitalized in HDJ Nutrition.

The results of this study will help confirm the association of muscle status on quality of life in obese patients, which is not yet clearly established in the scientific literature. If appropriate, these results will make it possible to propose non-invasive and inexpensive predictive tools to screen for muscle damage in this patient population. This screening could make it possible to propose early management programmes, such as exercise re-training or the introduction of adapted physical activity.

10. Expected benefits for the patient The use of non-invasive tests of muscle function could allow early identification of obese subjects whose impairment of muscle function could be associated with a poorer quality of life. This could allow us to propose an adapted therapeutic strategy, such as the implementation of an exercise training programme, adapted physical activity or therapeutic education.

ELIGIBILITY:
Inclusion Criteria:

Patients with the following criteria will be included:

* Outpatients assessment Nutrition ;
* Obese patients (BMI > 30);
* Patient at least 18 years old at the time of inclusion;
* Affiliation with a social security scheme or beneficiary of such a scheme ;
* Oral, free, informed and express consent of the patient.

Exclusion Criteria:

* Patient's refusal to participate in the study ;
* Known pregnancy ;
* Patient whose state of consciousness is not compatible with obtaining consent ;
* Person subject to a legal protection measure ;
* Patient under guardianship or curatorship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Outpatients assessment nutrition will be recruited prospectively and consecutively
Sampling Method: Probability Sample
Enrollment: 84 (Actual)
Dates: Start 2022-04-22 (Actual); Primary Completion 2023-07-22 (Actual); Study Completion 2023-10-02 (Actual)

PRIMARY OUTCOMES:
Association between structural alteration of the quadriceps and quality of life in obese patients | Through study completion, an average of 9 months
  The main outcome is the association between rectus femoris muscle echogenicity in the gray scale and the 36-Item Short Form Survey (SF-36) score

SECONDARY OUTCOMES:
The association between quadriceps thickness and quality of life | Through study completion, an average of 9 months
  The main outcome is the association between ultrasound thickness of the rectus femoris and the 36-Item Short Form Survey (SF-36) score
Association between grip strength and quality of life | Through study completion, an average of 9 months
  The main outcome is the association between grip strength measured by the hand-grip and the 36-Item Short Form Survey (SF-36) score
Association between quadriceps strength and quality of life | Through study completion, an average of 9 months
  The main outcome is the association between quadriceps maximal voluntary force on dynamometry and the 36-Item Short Form Survey (SF-36) score
Association between quadriceps strength and ultrasound measurements of the quadriceps | Through study completion, an average of 9 months
  The main outcome is the association between quadriceps FMV with dynamometry and ultrasound measurements of the rectus femoris (thickness, echogenicity and mCSA)

CONTACTS AND LOCATIONS:
Overall Officials: Sophie VIDAL-JESSEL, MD, Study Director — Hopital Forcilles; Andreia GOMES LOPES, MSc, Principal Investigator — Hopital Forcilles; Aymeric Le Neindre, PhD, Study Chair — Hopital Forcilles
Locations (1):
- Hôpital Forcilles, Férolles-Attilly, France

IPD SHARING:
Plan to Share IPD: Yes
The protocole, the statistical analysis plan and data will be available as supplementary materials with the publication. The other data that support the findings of this study will be available from the corresponding author upon reasonable request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: At publication for 10 years
Access Criteria: The data that support the findings of this study will be available from the corresponding author upon reasonable request.

REFERENCES:
- [Background] Toselli S, Campa F, Spiga F, Grigoletto A, Simonelli I, Gualdi-Russo E. The association between body composition and quality of life among elderly Italians. Endocrine. 2020 May;68(2):279-286. doi: 10.1007/s12020-019-02174-7. Epub 2019 Dec 31. PMID 31893349
- [Background] Tamura LS, Cazzo E, Chaim EA, Piedade SR. Influence of morbid obesity on physical capacity, knee-related symptoms and overall quality of life: A cross-sectional study. Rev Assoc Med Bras (1992). 2017 Feb;63(2):142-147. doi: 10.1590/1806-9282.63.02.142. PMID 28355375
- [Background] Kim SR, Kim HN, Song SW. Associations Between Mental Health, Quality of Life, and Obesity/Metabolic Risk Phenotypes. Metab Syndr Relat Disord. 2020 Sep;18(7):347-352. doi: 10.1089/met.2020.0028. Epub 2020 May 19. PMID 32429802

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2022-02-17): https://cdn.clinicaltrials.gov/large-docs/20/NCT05467020/Prot_SAP_ICF_000.pdf